CLINICAL TRIAL: NCT01327378
Title: The Incretin Effect in Non-diabetic Patients With Severe Renal Impairment Depending on Chronic Dialysis Treatment
Brief Title: The Incretin Effect in Patients With Kidney Impairment
Acronym: UREMINC
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Thomas Idorn/M.D. PhD student, Department of Nephrology, Rigshospitalet, University of Copenhagen, Denmark
Other Study IDs: H-C-2009-007
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2010-06

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma (10 ml per participant)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dialysis, normal glucose tolerance: Chronic dialysis treatment, N=10 OGTT,120 min < 7.8 mmol/L
- Dialysis, impaired glucose tolerance: Chronic dialysis treatment, N=10 OGTT,120 min 7.7<11.1 mmol/L
- Control, normal glucose tolerance: Healthy Control subjects, N=10 OGTT,120 min <7.8 mmol/L

SUMMARY:
The current study explores the incretin effect; a central mechanism of sugar metabolism. People with type 2 diabetes have a markedly reduced incretin effect, while the incretin effect never has been studied in patients with severe chronic renal failure. Non-diabetic patients with severe kidney failure and patients with diabetes and normal kidney function share several pathophysiological traits, including decreased sensitivity to insulin, fasting hyperinsulinaemia and impaired beta cell function. The investigators expect the incretin effect to be affected in patients with chronic renal failure without diabetes, which in time can result in therapeutic changes in this group of patients.

DETAILED DESCRIPTION:
The novel and original aspect of this investigator initiated study is the focus on incretin (patho)physiology in an uraemic milieu. In this first of 5 substudies (separate notification and registration) the investigators explore the incretin effect. Our hypothesis is that it is impaired in non-diabetic patients in chronic dialysis treatment.

The prevalence of type 2 diabetes mellitus (T2DM) is rapidly increasing worldwide. In addition to reduced insulin sensitivity and beta cell dysfunction, T2DM is characterized by a severely impaired incretin effect. The incretin effect refers to the insulinotropic action of the nutrient-released incretin hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP). Both hormones are secreted from intestinal endocrine mucosal cells. The incretin effect is defined as the difference in insulin secretory responses between oral and isoglycaemic intravenous (iv) glucose challenges. In healthy individuals it accounts for as much as 70% of insulin secreted in response to oral glucose, whereas patients with T2DM exhibit an incretin effect in the range of 0 to 30%. The incretin hormone GLP-1 has a potent blood glucose-lowering effect in patients with T2DM. However, following secretion of GLP-1, the ubiquitous enzyme dipeptidyl peptidase-4 (DPP-4) rapidly cleaves the hormone, by which it is completely inactivated. This has formed the basis for new pharmacological agents blocking DPP-4 (DPP-4 inhibitors) or DPP-4 resistant GLP-1 receptor agonists. Long-term treatment has showed positive effect on glycaemic control and risk factors of cardiovascular diseases in patients with T2DM.

These effects may be applicable also in patients with end-stage renal disease (ESRD) because patients with T2DM and normal kidney function and non-diabetic patients with ESRD show several identical characteristics. These include decreased insulin sensitivity, hyperinsulinaemia and impaired beta cell function. The incretin effect has only to a small extent been investigated in patients with ESRD.

The single most frequent cause of ESRD and need of chronic maintenance dialysis is diabetic nephropathy. In the U.S. more than 50% of patients in dialysis have diabetes compared with about 23% in Denmark. The life expectancy of dialysis patients with T2DM is severely reduced with a median survival of 2 to 4 years and there is no treatment documented to significantly improve this poor prognosis. The most common cause of death in this group of patients is related to cardiovascular disease that seems to result from death of causes different from classical atherosclerosis. So far intervention directed towards hypertension, dyslipidaemia and other classical risk factors have showed divergent and primarily negative results.

There is therefore an unmet medical need to find new treatments to protect these patients from cardiovascular disease and premature death.

Improving the glycaemic control using incretin-based therapies has the potential to meet this medical need. The incretin hormones and their metabolites are however to a large extent excreted by the kidneys and this may lead to problems (or benefits!) when administered to patients without kidney function or with severely reduced kidney function. The present knowledge about the incretin effect and incretin hormone physiology as well as pharmacokinetics, clinical effects and side effects of GLP-1 analogues in patients with reduced kidney function is limited and the few studies available are predominantly confined to patients with only mild or moderately reduced kidney function. The investigators will explorer basic and pharmacologic aspects in patients with severe reduced kidney function depending on chronic maintenance dialysis treatment. Before any potential treatment can be initiated, the investigators need basic information on how the incretin system is affected by an uraemic milieu. Current and succeeding substudies will provide us with that information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age: 18 - 90 years
* CKD stage 5 (CrCL < 15 ml/min) in chronic haemodialysis (minimum 3 months)
* NGT or IGT (diagnosed according to WHO criteria)
* Body mass index 18.5 - 28 kg/m2

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Pancreatitis
* Medication with influence on insulin secretion and/or glucose metabolism
* Previous or actual malignancy
* Inflammatory bowel disease
* Congestive heart failure (NYHA III-IV)
* Previous bowel resection
* Severe hypertension
* Impaired liver function
* Haemoglobin < 6.5 mmol/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups
  1. Chronic hemodialysis treatment. Normal glucose tolerance (NGT). N=10
  2. Chronic hemodialysis treatment. Impaired glucose tolerance (IGT). N=10
  3. Healthy control subjects. Normal glucose tolerance. N=10
  Glucose tolerance is evaluated at the screeningday. A 75 gram oral glucose tolerance test (OGTT) is performed and the 120 minute value sets the glucose tolerance. NGT: < 7.8 mmol/L, IGT: > 7.7 mmol/L and < 11.1 mmol/L (according to WHO guidelines).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incretin effect | Minimum 3 days and maximum 3 weeks between the two examination days. Cross-sectional design. No follow up.
  IE= 100%*(iAUC,OGTT - iAUC,IIGI)/iAUC,OGTT Assessed at two separate examination days. Day 1: Oral glucose tolerance test (OGTT), Day 2: Intravenous isoglycaemic glucose infusion (IIGI).
  Data will be presented when all analyses have been performed. Estimated in May 2011.

SECONDARY OUTCOMES:
Gastric-induced glucose disposal (GIGD) | Minimum 3 days and maximum 3 weeks between the two examination days. Cross-sectional design. No follow up.
  GIGD=100%*(glucose,OGTT-glucose,IIGI)/glucose,OGTT) Assessed at two separate examination days. Day 1: Oral glucose tolerance test (OGTT), Day 2: Intravenous isoglycaemic glucose infusion (IIGI).
  Data will be presented when all analyses have been performed. Estimated in May 2011.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Prof, DMSc, Study Director — Department of Nephrology, Rigshospitalet, University of Copenhagen, Denmark
Locations (1):
- Department of Nephrology P 2131, Rigshospitalet, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Wewer Albrechtsen NJ, Hartmann B, Veedfald S, Windelov JA, Plamboeck A, Bojsen-Moller KN, Idorn T, Feldt-Rasmussen B, Knop FK, Vilsboll T, Madsbad S, Deacon CF, Holst JJ. Hyperglucagonaemia analysed by glucagon sandwich ELISA: nonspecific interference or truly elevated levels? Diabetologia. 2014 Sep;57(9):1919-26. doi: 10.1007/s00125-014-3283-z. Epub 2014 Jun 3. PMID 24891019
- [Derived] Idorn T, Knop FK, Jorgensen M, Holst JJ, Hornum M, Feldt-Rasmussen B. Gastrointestinal factors contribute to glucometabolic disturbances in nondiabetic patients with end-stage renal disease. Kidney Int. 2013 May;83(5):915-23. doi: 10.1038/ki.2012.460. Epub 2013 Jan 16. PMID 23325073